CLINICAL TRIAL: NCT04385446
Title: Comparative Study of Concentration of Muc5ac and Muc2 Mucins in Tear Film in Surgical Treated Pterygia With Amniotic Membrane Transplantation vs. Conjunctival Autograft
Brief Title: Comparative Study of Muc5ac and Muc2 Mucins in Tear Film Concentration in Surgical Treated Pterygia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: CC-001/105
Record Dates: First submitted 2020-04-29; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-04

CONDITIONS: Pterygium of Both Eyes
Keywords: pterygium, amniotic membrane, conjunctival autograft, ocular mucin
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Intervention Model Description: Two groups of patients in whom Conventional Pterygium surgery was performed Each patient was randomly assigned for either received amniotic membrane transplantation or conjunctival autograft as a recovering method in the pterygium removed area after surgery. Tear film Mucins were measured in both groups
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients did not know what kind of material was used in their surgery. The assessor who performed tear film analysis did not know what material was used in the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amniotic membrane transplantation (Active Comparator): Amniotic membrane transplantation was used as covering material in the area where the pterygium tissue was removed during the surgery.
  Interventions: Procedure: Amniotic membrane transplantation
- conjnctival autograft. (No Intervention): Conjunctival autograft was used as a covering material in the area where the pterygium tissue was removed during the surgery.

INTERVENTIONS:
Procedure: Amniotic membrane transplantation — Amniotic membrane transplantation was used as covering material during pterygium surgery.
  Arms: Amniotic membrane transplantation

SUMMARY:
To identify and compare the differences in the concentration of the Muc2 and Muc5AC mucins in tear film in patients who underwent pterygium surgery using amniotic membrane transplantation and conjunctival autograft surgery.

DETAILED DESCRIPTION:
Patients with nasal, primary pterygium bigger than 1 mm of corneal invasion with residence in Mexico City and older than 18 years were included. Under informed consent, patients were divided into two groups in a random fashion. Pterygium surgery was carried out with conventional technique performing amniotic membrane transplantation for group A, and conjunctival autograft for group B. Muc2 and muc5ac mucin concentration was measure min tear film by ELISA; samples were taken before surgery, at first, third and sixth month postoperatively. BUT was also measured on the same dates. Descriptive statistics and the U-Mann Whitney test for independent groups, considering a p≤0.05 as significant were used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with nasal, primary pterygium bigger than 1 mm.

Exclusion Criteria:

* Diabetes mellitus, single eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2017-02-07 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
Ocular Tear film Mucin MUC5ac concentration. | The patients will be assed during six months
  Using a capillary tube, tear film was collected en every patient. Then Concentration of mucin MUC5ac were measured by Elisa technique using a quantitative scale.
Ocular tear film Mucin MUC2 concentration. | The patients will be assed during six months
  Using a capillary tube, tear film was collected en every patient. Then Concentration of mucin MUC2 were measured by Elisa technique using a quantitative scale.
Tear film breakup time. | The patients will be assed during six months
  Tear film breakup time is the time between a complete blink and the appearance of the first random corneal dry spot and indicates relative tear film stability.

SECONDARY OUTCOMES:
Pterygium recurrence. | The patients will be assed during six months
  Pterygium recurrence was defined as any fibrovascular proliferation from the original pterygium site from it was surgically removed.